CLINICAL TRIAL: NCT00014937
Title: A Randomized, Controlled Trial of Two Potent, Simplified Regimens Utilizing A Protease Inhibitor-Sparing Regimen Versus A Nucleoside-Sparing Regimen for HIV-Infected Subjects Who Participated in ACTG 388 or Who Responded to A First Potent Combination Regimen and Have 200 or Less HIV-1 RNA Copies/ml
Brief Title: Simplified Drug Regimens for HIV Patients in ACTG 388 or Patients Who Responded to A First Potent Combination Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: A5116; AACTG 5116; Substudy AACTG A5124s; Substudy AACTG A5125s; ACTG A5116; 10934 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2001-04-14; First posted 2001-08-31 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Didanosine; Drug Therapy, Combination; Zidovudine; Nevirapine; Stavudine; HIV Protease Inhibitors; Ritonavir; Lamivudine; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; ABT 378; Combivir; Efavirenz; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; lamivudine, zidovudine drug combination; efavirenz; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: lopinavir/ritonavir
Drug: lamivudine/zidovudine
Drug: efavirenz
Drug: lamivudine
Drug: stavudine
Drug: zidovudine
Drug: didanosine

SUMMARY:
ACTG 388 was a clinical trial that compared three- and four-drug anti-HIV drug regimens and demonstrated the effectiveness of a three-drug regimen. This study will compare the ability of two different three-drug anti-HIV drug regimens to reduce levels of HIV in the blood. The study will also evaluate whether patients discontinue the regimens because of drug side effects.

DETAILED DESCRIPTION:
ACTG 388 was designed to evaluate two four-drug regimens compared with a three-drug regimen in patients who were relatively treatment naive. Based on the increased complexity and toxicity of four-drug regimens and the resultant negative impact on response as compared with three-drug regimens, studies evaluating simplified potent regimens appear warranted. This study will evaluate simpilified drug regimens designed to enhance virologic activity without necessarily increasing the number of antiretroviral drugs. The study regimens will be assessed for both virologic control and tolerability. The study population will include patients previously enrolled in ACTG 388 and patients with prior advanced HIV disease who received and responded to potent antiretroviral therapy without evidence of virologic relapse.

Patients will be stratified according to ACTG 388 treatment or non-ACTG 388 study participation. Patients will then be randomized to receive either a protease inhibitor (PI)-sparing regimen of 2 nucleoside reverse transcriptase inhibitors (NRTIs) with efavirenz (EFV) (Arm I) or an NRTI-sparing regimen of EFV with lopinavir/ritonavir (LPV/r) (Arm II). Arm I options are enteric-coated didanosine (ddI-EC) plus lamivudine (3TC), ddI-EC plus zidovudine (ZDV), ZDV plus 3TC (or Combivir), stavudine (d4T) plus 3TC, or ddI-EC plus d4T (with exceptions as noted in the protocol). Only LPV/r, EFV, d4T, and ddI are provided by the study; other medications are obtained by nonstudy prescription.

All patients are evaluated for safety and for virologic and immunologic responses at Weeks 4 and 8, then every 8 weeks until the study ends. In addition, all patients have assessments for fat redistribution, fasting lipid profiles, fasting insulin levels, venous lactate levels, and treatment adherence. Patients will be followed for 1.5 to 3 years. Interim safety analyses will be conducted in June 2002 and June 2003. Patients in this study may also enroll in A5125s, a fat distribution and bone mineral density substudy.

ELIGIBILITY:
Inclusion Criteria for ACTG 388 Participants

* HIV-1 RNA level <= 200 copies/ml within 70 days of study entry
* Stable anti-HIV drug plan without harmful drug side effects or serious illness at the time of study entry

Inclusion Criteria for Non-ACTG 388 Participants

* Potent anti-HIV drug regimen as a first HIV treatment for at least 18 months
* HIV-1 RNA level >= 80,000 copies/ml or CD4+ count <= 200 cells/mm3 prior to starting anti-HIV drug regimen
* HIV-1 RNA level <= 400 copies/ml (or less than 500 copies/ml by bDNA) within 32 weeks of initial therapy
* HIV-1 RNA level <= 200 copies/ml within 60 days of study entry

Inclusion Criteria for Both ACTG 388 and Non-ACTG 388 Participants

* Acceptable methods of contraception
* Consent of parent or legal guardian if under 18 years of age

Exclusion Criteria for ACTG 388 Participants

* Viral resistance to study drugs as determined by resistance studies during ACTG 388

Exclusion Criteria for ACTG 388 and Non-ACTG 388 Participants

* Pregnancy or breastfeeding
* Certain heart medicines (flecainide or propafenone); antihistamines (astemizole and terfenadine); rifampin; ergot derivatives (dihydroergotamine, ergonovine, ergotamine, or methylergonovine); intestinal agents (cisapride); herbal products (St. John's wort); lovastatin or simvastatin; neuroleptics (pimozide); and sedatives/hypnotics (midazolam or triazolam)
* Allergy study drugs

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Fischl, MD, Study Chair — University of Miami
Locations (37):
- United States (32):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Denver Dept of Health and Hosps, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Connecticut Children's Medical Center (Pediatric), Farmington, Connecticut
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Univ of Minnesota, Minneapolis, Minnesota
  - Washington Univ / St Louis Connect Care, St Louis, Missouri
  - Washington Univ School of Medicine, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Washington, Seattle, Washington
- Italy (4):
  - Spedali Civili - Carosi, Brescia
  - Universita di Genova, Genova
  - Ospedale Luigi Sacco Milazzo, Milan
  - Universita degli Studi di Modena e Reggio Emilia, Modena
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Demeter LM, Ribaudo HJ, Erice A, Eshleman SH, Hammer SM, Hellmann NS, Fischl MA; AIDS Clinical Trials Group Protocol 388. HIV-1 drug resistance in subjects with advanced HIV-1 infection in whom antiretroviral combination therapy is failing: a substudy of AIDS Clinical Trials Group Protocol 388. Clin Infect Dis. 2004 Aug 15;39(4):552-8. doi: 10.1086/422518. Epub 2004 Jul 30. PMID 15356820
- [Result] Tebas P, Zhang J, Yarasheski K, Evans S, Fischl MA, Shevitz A, Feinberg J, Collier AC, Shikuma C, Brizz B, Sattler F; AIDS Clinical Trials Group (ACTG). Switching to a protease inhibitor-containing, nucleoside-sparing regimen (lopinavir/ritonavir plus efavirenz) increases limb fat but raises serum lipid levels: results of a prospective randomized trial (AIDS clinical trial group 5125s). J Acquir Immune Defic Syndr. 2007 Jun 1;45(2):193-200. doi: 10.1097/QAI.0b013e318042e204. PMID 17527093